CLINICAL TRIAL: NCT05997537
Title: Dynamic Web-Based Interventions to Improve Update of Preventive Health Recommendations in IBD
Status: Completed | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Gil Melmed, Clinical Director of Inflammatory Bowel Disease, Cedars-Sinai Medical Center
Other Study IDs: Pro00056067
Record Dates: First submitted 2023-08-04; First posted 2023-08-18 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: IBD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To understand patient knowledge, attitudes, and beliefs around the uptake of vaccinations and malignancy screening through patient focus groups/qualitative interviews. To develop and pilot an interactive website that will provide customized recommendations for individual patients with IBD and direct them as relevant to five 60-90 second customized, animated videos (influenza, pneumococcal, and zoster vaccinations, bone health, and skin cancer screening). This content will be pilot-tested with patients to fine-tune the educational modules.

ELIGIBILITY:
Inclusion Criteria:

* enrollees in the internet-based cohort IBD Partners, age 18 and older

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled in IBD Partners, age 18 and older who have agreed to be contacted for future studies.
Sampling Method: Probability Sample
Enrollment: 1056 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-03-07 (Actual)

PRIMARY OUTCOMES:
Uptake of influenza vaccination | Through study completion, no later than March 31, 2020
  Uptake of influenza vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Gil Melmed, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai, Los Angeles, California, United States

REFERENCES:
- [Derived] Long MD, van Deen WK, Weisbein L, Khalil C, Appel KL, Zhang X, Chen W, Zubrod L, Maris R, Ghafari A, Dupuy T, Ha CY, Spiegel BMR, Almario CV, Melmed GY. Web-Based Video Education to Improve Uptake of Influenza Vaccination and Other Preventive Health Recommendations in Adults With Inflammatory Bowel Disease: Randomized Controlled Trial of Project PREVENT. J Med Internet Res. 2023 Aug 23;25:e42921. doi: 10.2196/42921. PMID 37610821